CLINICAL TRIAL: NCT06956040
Title: Involvement of General Practitioners in Lung Cancer Screening
Acronym: GEDEPIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230811; 2024-A00669-38 (Other: ID-RCB)
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: Screening; Lung cancer; General practitioners; CT Scan
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Low-dose computed tomography of the chest — Baseline low dose Ct acquisition, then at 1 year to depict suspicious lung nodules

SUMMARY:
The main objective is to evaluate the adherence of smoking patients to lung cancer screening by low-dose CT scan, when proposed by the general practitioner.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer mortality in France and worldwide. The KBP2020 study conducted in general hospitals, including 8999 patients diagnosed with lung cancer in the year 2020, showed that 73% of lung cancer cases were diagnosed at an advanced symptomatic stage, explaining the high rate of metastatic status at diagnosis, reaching 58%. For this category of patients, 3-month mortality remains very high, close to 25%. Several large randomized studies have demonstrated that lung cancer screening with low-dose CT scans enables lung cancer to be diagnosed at an early, asymptomatic stage, when it is mostly accessible to curative surgical treatment. This early detection and subsequent treatment reduced specific mortality by 20% in the NLST study, and by up to 39% at 10 years in the MILD study. Overall mortality was reduced by 6.7% in the NLST study. This scientific evidence has led the French National Authority for Health to encourage the implementation of a pilot program, to be organized by the French National Cancer Institute.

The hypothesis of the study is that the proposal of CT screening for lung cancer will be better adhered to if it is made by the general practitioner of individuals at risk. Adherence is defined by an initial scan, followed by a second scan one year after the first, with participation in screening on an annual basis.

Given the trust that generally characterizes the relationship between patients and their GP, and the fact that intercurrent consultations provide reminders of the need for an annual check-up, the assumption is for an initial participation rate of at least 50%, and a continued participation rate of 70% at 1 year.

Communication of results by the GP will help to limit anxiety, particularly in the event of an undetermined result, which will be assessed by the anxiety section of the Hospital Anxiety and Depression scale questionnaire translated into French.

In addition, the success of smoking cessation will be compared with literature data in the context of screening. The hypothesis is that the cessation rate will be higher due to the possibility of adapting nicotine substitution by the GP and his or her repeated support in the cessation process.

Finally, knowledge of patients' histories will help to limit unnecessary explorations and to better identify for which participants screening reveals COPD (emphysema), osteoporosis or unrecognized coronary artery disease.

ELIGIBILITY:
Inclusion Criteria :

* Adults aged 50-74
* Active smoker or weaned smoker for less than 15 years, of at least 20 pack-years
* Affiliation with a social security scheme or CMU (beneficiary or beneficiary entitled)
* Written informed consent prior to study participation

Exclusion Criteria :

* History of lung cancer
* Thoracic CT scan performed within the previous year
* 1-year follow-up not possible
* Inability to travel independently to Hôpital Cochin or Hôpital Bichat for scans
* People with severe co-morbidities contraindicating exploration and/or management of lung cancers
* People in poor general health (=PS2 and above)
* People with a history of cancer under active surveillance by thoracic computed tomography (CT and PET scans)
* People with rest dyspnea (=mMRC4)
* Recent weight loss, altered general condition or hemoptysis, raising suspicion of progressive lung cancer
* Signs of respiratory infection (fever, productive cough)
* Patients under guardianship, curatorship or protected adults
* Inability to give free written informed consent prior to study participation

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of completion of screening scan | 12 months
  Rate of completion of screening scan, one year after initial scan.

SECONDARY OUTCOMES:
Evolution of tobacco consumption | 12 months
  Comparison of tobacco consumption at 1 year versus consumption at baseline
Evolution of anxiety | 12 months
  Hospital Anxiety and Depression Scale score (anxiety section) completed by the participant at the initial scan, at 1 year (and any additional scans), at follow-up consultations with the GP (and any additional scans) and at the end of the study.
  The minimum score is 0 and the maximum is 21. Higher score means worse outcome.
Chronic obstructive pulmonary disease (COPD) | Up to 12 months
  Number of participants with initially unrecognized COPD confirmed by lung function tests.
Statin/aspirin prevention | Up to 12 months.
  Number of participants for whom statin/aspirin prevention is initiated following initial scan.
Osteoporosis | Up to 12 months.
  Number of participants with osteoporosis not known at inclusion confirmed by bone densitometry.
Other pathologies | Up to 18 months
  Number of other pathologies confirmed by their reference examination.
Cancer screened | Up to 18 months
  Rate of stage I cancers among screened cancers.
Characteristics of eligible population refusing screening : age | Day 0
  Age of eligible people refusing screening
Characteristics of eligible population refusing screening : sex | Day 0
  Sex of eligible people refusing screening
Characteristics of eligible population refusing screening : smoking status | Day 0
  Smoking status of eligible people refusing screening
Characteristics of eligible population refusing screening : level of education | Day 0
  Level of education of eligible people refusing screening
Characteristics of eligible population refusing screening : reason for refusal | Day 0
  Reason for refusal of eligible people refusing screening

CONTACTS AND LOCATIONS:
Overall Officials: Céline BUFFEL du VAURE, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marie-Pierre REVEL, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Christian GHASAROSSIAN, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosell R, Gonzalez-Cao M. Ablating lung cancer, knowing the tumor better. Lancet Reg Health Eur. 2022 Aug 26;22:100494. doi: 10.1016/j.lanepe.2022.100494. eCollection 2022 Nov. No abstract available. PMID 36061495
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Pastorino U, Silva M, Sestini S, Sabia F, Boeri M, Cantarutti A, Sverzellati N, Sozzi G, Corrao G, Marchiano A. Prolonged lung cancer screening reduced 10-year mortality in the MILD trial: new confirmation of lung cancer screening efficacy. Ann Oncol. 2019 Jul 1;30(7):1162-1169. doi: 10.1093/annonc/mdz117. PMID 30937431
- [Background] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683
- [Background] Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, Padonu G, Talarczyk G. Patient satisfaction with health care decisions: the satisfaction with decision scale. Med Decis Making. 1996 Jan-Mar;16(1):58-64. doi: 10.1177/0272989X9601600114. PMID 8717600
- [Background] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Hussain MS, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. AJNR Am J Neuroradiol. 2018 Jun;39(6):E61-E76. doi: 10.3174/ajnr.A5638. Epub 2018 May 17. No abstract available. PMID 29773566
- [Background] Leleu O, Basille D, Auquier M, Clarot C, Hoguet E, Baud M, Lenel S, Milleron B, Berna P, Jounieaux V. Results of Second Round Lung Cancer Screening by Low-Dose CT scan - French Cohort Study (DEP-KP80). Clin Lung Cancer. 2022 Jan;23(1):e54-e59. doi: 10.1016/j.cllc.2021.09.009. Epub 2021 Oct 10. PMID 34764039
- [Background] Aubin-Auger I, Laouenan C, Le Bel J, Mercier A, Baruch D, Lebeau JP, Youssefian A, Le Trung T, Peremans L, Van Royen P. Efficacy of communication skills training on colorectal cancer screening by GPs: a cluster randomised controlled trial. Eur J Cancer Care (Engl). 2016 Jan;25(1):18-26. doi: 10.1111/ecc.12310. Epub 2015 Apr 6. PMID 25851842
- [Background] Aim-Eusebi A, Cussac F, Aubin-Auger I. [Cancer prevention and screening: What french GPs could do?]. Bull Cancer. 2019 Jul-Aug;106(7-8):707-713. doi: 10.1016/j.bulcan.2018.11.015. Epub 2019 Jan 17. French. PMID 30661748
- [Background] Custers JA, van den Berg SW, van Laarhoven HW, Bleiker EM, Gielissen MF, Prins JB. The Cancer Worry Scale: detecting fear of recurrence in breast cancer survivors. Cancer Nurs. 2014 Jan-Feb;37(1):E44-50. doi: 10.1097/NCC.0b013e3182813a17. PMID 23448956
- [Background] Shemesh J, Henschke CI, Shaham D, Yip R, Farooqi AO, Cham MD, McCauley DI, Chen M, Smith JP, Libby DM, Pasmantier MW, Yankelevitz DF. Ordinal scoring of coronary artery calcifications on low-dose CT scans of the chest is predictive of death from cardiovascular disease. Radiology. 2010 Nov;257(2):541-8. doi: 10.1148/radiol.10100383. Epub 2010 Sep 9. PMID 20829542